CLINICAL TRIAL: NCT00486083
Title: A Randomized, Double-Blind Comparison, Safety and Efficacy Trial of Atomoxetine Hydrochloride and Methylphenidate Hydrochloride in Pediatric Outpatients With DSM-IV Attention-Deficit/Hyperactivity Disorder
Brief Title: Comparison Atomoxetine Hydrochloride and Comparator in Pediatric Outpatients With ADHD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 6934; B4Z-MC-LYBR
Record Dates: First submitted 2007-06-11; First posted 2007-06-13 (Estimated); Last update posted 2007-06-13 (Estimated); Status verified 2007-06

CONDITIONS: Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Atomoxetine Hydrochloride; Methylphenidate

INTERVENTIONS:
Drug: Atomoxetine Hydrochloride
Drug: Methylphenidate Hydrochloride

SUMMARY:
The purpose of the study is to compare atomoxetine hydrochloride and methylphenidate hydrochloride in pediatric patients with ADHD.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 6 years of age and not more than 16 years of age at Visit 1
* Must meet DSM-IV criteria for ADHD
* Must be of normal intelligence (that is, without a general impairment of intelligence and likely, in the investigator's judgement, to achieve a score of greater than or equal to 70 on an IQ test)
* Must be able to swallow capsules
* Must have laboratory results that show no significant abnormalities (significant would include laboratory deviations requiring acute medical intervention or further medical evaluation)

Exclusion Criteria:

* Weigh less than 20 kg or more than 60 kg at study entry
* Have a history of Bipolar I or II disorder, psychosis, or pervasive developmental disorder
* Meet DSM-IV criteria for an anxiety disorder
* Have a history of any seizure disorder (other than febrile seizures)or prior ECG abnormalities related to epilepsy, or subjects who have taken or are currently taking anti-convulsants for seizure control
* Have a history of severe allergies to more than 1 class of medications or multiple adverse drug reactions,including a hypersensitivity to methylphenidate

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 330 (Actual)
Dates: Start 2003-12; Study Completion 2004-10 (Actual)

PRIMARY OUTCOMES:
Test the hypothesis that atomoxetine hydrochloride is non-inferior to methylphenidate hydrochloride in improving ADHD symptoms following an approximately 8-week period of double blind treatment as assessed by a comparison of response rates

SECONDARY OUTCOMES:
To compare the tolerability of atomoxetine and methylphenidate as assessed by treatment-emergent adverse events
To assess the comparability of the efficacy of atomoxetine and methylphenidate on the Conners' Parent Rating Scale-Revised: Short Form
To compare atomoxetine and methylphenidate on other secondary measures

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (3):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Shanghai, China
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mexico City, Mexico
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seoul, South Korea

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com